CLINICAL TRIAL: NCT02501187
Title: Comparison Between Three Different Surgeries for Blepharoptosis Repair and Their Impact on Dry Eye Status
Brief Title: Risk of Dry Eye Post Different Surgeries for Blepharoptosis Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Maya Eiger, Medical Doctor, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ptosis-01
Record Dates: First submitted 2015-07-12; First posted 2015-07-17 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients operated for ptosis by levator advancement (Experimental): patients undergoing surgical repair for aponeurotic ptosis by the procedure- levator advancement.
  Interventions: Procedure: Levator advancement
- Patients operated for ptosis by white line advancement (Experimental): patients undergoing surgical repair for aponeurotic ptosis by the procedure- white line advancement
  Interventions: Procedure: White line advancement
- Patients operated for ptosis by Müller resection (Experimental): patients undergoing surgical repair for aponeurotic ptosis by the procedure- Müller's muscle-conjunctival resection.
  Interventions: Procedure: Müller's muscle-conjunctival resection procedure

INTERVENTIONS:
Procedure: Levator advancement — A transcutaneous procedure in which the Levator palpebrae aponeurosis is advanced and attached to the tarsus.
  Arms: Patients operated for ptosis by levator advancement
Procedure: Müller's muscle-conjunctival resection procedure — A transconjunctival procedure in which part of the muller muscle and conjunctiva are resected.
  Arms: Patients operated for ptosis by Müller resection
Procedure: White line advancement — A transconjunctival procedure in which the Levator palpebrae aponeurosis is advanced and attached to the tarsus.
  Arms: Patients operated for ptosis by white line advancement

SUMMARY:
Blepharoptosis, inferodisplacement of the upper eyelid, can be congenital or acquired. Acquired Blepharoptosis is usually aponeurotic, due to stretching or disinsertion of the levator aponeurosis. Treatment is surgical and can be performed by three common procedures - Levator advancement, Müller's muscle-conjunctival resection procedure and White line advancement. A number of reports inspected the possibility that Blepharoptosis repair procedures may cause deterioration in dry eye status. The investigators would like to assess whether there is a difference between the different procedures in their influence on dry eye status.

ELIGIBILITY:
Inclusion Criteria:

* Ptosis which indicate surgical repair
* The ptosis must be suitable for repair in any of the procedures

Exclusion Criteria:

* Systemic disease which may cause ocular surface disease (eg Sjogren disease)
* Previous orbital or eyelid surgery
* Significantly dry eyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-10-08 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of objective or subjective deterioration in dry eye status | 6 months
  Dry eye status will be measured by a composite of tests, including Ocular surface disease index (OSDI) questionnaire (which indicates subjective status), and a number of objective tests - Shirmer test, Flurocein dye, Lissamine green dye and tear breakup time

SECONDARY OUTCOMES:
Ptosis repair procedure success | 6 months
  Success will be assessed by comparison of margin reflex distance1 (MRD1) measurement before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maya Eiger, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Ophthalmology clinics, Rabin Medical Center, Petah Tikva, Israel